CLINICAL TRIAL: NCT06205615
Title: Randomized, Double-Blind, Placebo-Controlled, 2-Way Crossover Study to Evaluate the Efficacy and Safety of BXP154B (Tranexamic Acid Sterile Topical Solution) in the Treatment of External Bleeding From Minor Wounds in Subjects on Apixaban
Brief Title: Treatment of Post-Punch Biopsy Bleeding in Apixaban-Treated Patients Using Self-Administered BXP154B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bio 54, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BXP154-201
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Wound Bleeding
Keywords: Anticoagulant

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, 2-way crossover
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Punch Biopsy + BXP154B/Right Leg Period 1; Punch Biopsy + Placebo/Left Leg Period 2 (Experimental): Single topical application of BXP154B 6ml after punch biopsy (right leg), treatment period 1; single topical application of Placebo 6ml after punch biopsy (left leg), treatment period 2
  Interventions: Drug: BXP154B; Drug: Placebo; Procedure: Punch Biopsy
- Punch Biopsy + Placebo/Right Leg Period 1; Punch Biopsy + BXP154B/Left Leg Period 2 (Experimental): Single topical application of Placebo 6ml after punch biopsy (right leg), treatment period 1; single topical application of BXP154B 6ml after punch biopsy (left leg), treatment period 2
  Interventions: Drug: BXP154B; Drug: Placebo; Procedure: Punch Biopsy
- Punch Biopsy + BXP154B/Left Leg Period 1; Punch Biopsy + Placebo/Right Leg Period 2 (Experimental): Single topical application of BXP154B 6ml after punch biopsy (left leg), treatment period 1; single topical application of Placebo 6ml after punch biopsy (right leg), treatment period 2
  Interventions: Drug: BXP154B; Drug: Placebo; Procedure: Punch Biopsy
- Punch Biopsy + Placebo/Left Leg Period 1; Punch Biopsy + BXP154B/Right Leg Period 2 (Experimental): Single topical application of Placebo 6ml after punch biopsy (left leg), treatment period 1; single topical application of BXP154B 6ml after punch biopsy (right leg), treatment period 2
  Interventions: Drug: BXP154B; Drug: Placebo; Procedure: Punch Biopsy

INTERVENTIONS:
Drug: BXP154B — BXP154B will be self-administered topically following wound induction
Drug: Placebo — Placebo will be self-administered topically following wound induction
Procedure: Punch Biopsy — Punch biopsy to leg

SUMMARY:
The goal of this clinical trial is to test if the study drug, BXP154B works to stop bleeding from a minor wound in patients that are on apixaban for anticoagulant therapy. The main questions it aims to answer are:

* How long does it take to stop bleeding after BXP154B is applied to a wound?
* How many people require the use of a rescue treatment to stop bleeding?
* Does BXP154B reduce instances of re-bleeding after the bleeding has stopped initially?
* Is BXP154B safe and well-tolerated?

DETAILED DESCRIPTION:
Oral anticoagulant-related clinically relevant nonmajor bleeding (CRNMB; i.e., non-major bleeding that requires medical intervention, increased level of care, or face-to-face evaluation) and minor bleeding, often referred to as 'nuisance' bleeding, carries a high burden in terms of patient discomfort, anxiety, temporary disability, and reduced quality of life, and strain on medical and socioeconomic resources. Prolonged bleeding following minor injuries (falls, scrapes, cuts) can be life-interrupting and frequently leads patients to seek medical care, often times in an urgent care or emergency department (ED) setting. Prolonged bleeding from minor injuries is a significant challenge to daily life for people on anticoagulants, and is anything but 'minor' to the patient.

Bio 54, LLC, is developing BXP154B, a topical agent intended for self-administration (in or outside the home) to treat external bleeding from minor wounds in patients on anticoagulants. The development of BXP154B will offer patients on anticoagulants a much-needed treatment for self-management of external bleeding from minor wounds at home.

BXP154-201 is a randomized, double-blind, placebo-controlled, 2-way crossover-design study to evaluate the efficacy and safety of BXP154B (6 mL) compared with volume-matched placebo in the treatment of bleeding following punch biopsy in subjects on apixaban.

Subjects will be enrolled in this clinical trial for a total of seven days, following a screening period of up to 28 days. The study commences on Day 1 with a skin punch biopsy and administration of the investigational drug or placebo. Subsequently, follow-up assessments will be conducted on Days 2, 3, and 4. A second skin punch biopsy will be performed on Day 4, followed by additional follow-up assessments on Days 5, 6, and 7. Upon completion of the Day 7 assessments, subjects will have fulfilled their involvement in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age on the day of signed informed consent. At least 8 subjects of each sex will be enrolled.
* Currently receiving apixaban (Eliquis®) and on a BID dosing regimen 5 mg BID (10 mg total daily dose). Subjects must have been on the same dosing regimen for at least 7 days prior to Day 1.
* Willing and able to provide informed consent prior to any study procedures and to comply with all aspects of the protocol

Exclusion Criteria:

* Allergy or sensitization to any components of BXP154B
* BMI ≥ 50 kg/m2
* Known genetic/familial hypercoagulable disorder
* Thrombocytopenia (platelets <75,000/mm3)
* Subjects using any prescribed chronic drug therapies that impact platelet function including clopidogrel (Plavix®), prasugrel (Effient®), ticagrelor (Brillinta®), dipyridamole (Aggrenox®), cilostazol (Pletal®), aspirin, or any non-steroidal anti-inflammatory drugs (NSAIDs; e.g., ibuprofen, naproxen, diclofenac, indomethacin, ketorolac, etc.) are excluded from participation in the study. NSAIDs or aspirin taken on an as needed (PRN) basis must be discontinued according to the following required windows prior to Day 1 (aspirin, 7 days; ibuprofen, 24 hours; all other NSAIDs, 4 days) and may not be taken for the duration of the study.
* Use of any other anticoagulant therapies other than apixaban 5mg BID
* Hypersensitivity to any local anesthetic being used by the site
* Pregnant, breastfeeding, or planning to become pregnant
* Use of any hormonal contraceptive methods (e.g., oral, injectable, vaginal ring, transdermal patch, or hormonal intrauterine device [IUD]), or any oral treatment containing estrogen or synthetic estrogen within 30 days prior to Screening or during study participation. Women of childbearing potential must agree to use effective non-hormonal contraception during study participation.
* Participation in another clinical trial for an investigational product within 30 days prior to Screening. In addition, subjects who participated in BXP154-PIL are not eligible for this study.
* Any clinically significant finding on screening assessments or other physical or neurological condition that, in the opinion of the investigator, impairs the ability of the subject to comply with protocol procedures and safely participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Time to achieve hemostasis (in minutes) following start of treatment | 60 minutes following start of treatment
  Time to achieve hemostasis (in minutes) will be compared between active treatment and control.

SECONDARY OUTCOMES:
Proportion of subjects who achieve hemostasis within 4mins, 8mins, 12mins, 16mins, 20mins, 25mins, 30mins, 40 mins, 50mins, 60mins | 60 minutes following start of treatment
  Summarized as the proportion of subjects that met criteria and compared between active treatment and control.
Proportion of subjects who require rescue treatment intervention to achieve hemostasis following biopsy | 60 minutes following start of treatment
  Summarized as the proportion of subjects that met criteria and compared between active treatment and control.
Time to achieve hemostasis (in minutes) with no rebleeding requiring self-managed or medical intervention within 72 hours after the start of treatment | 72 hours following start of treatment
  Time (in minutes) to achieve hemostasis will be compared between active treatment and control.
Proportion of subjects who experience rebleeding following initial hemostasis that requires self-managed or medical intervention to re-achieve hemostasis within 24, 48, and 72 hours after the start of treatment | 72 hours following start of treatment
  Summarized as the proportion of subjects that met criteria and compared between active treatment and control.
Proportion of subjects who experience rebleeding following initial hemostasis that requires subsequent self-managed intervention to re-achieve hemostasis within 24, 48, and 72 hours after the start of treatment | 72 hours following start of treatment
  Summarized as the proportion of subjects that met criteria and compared between active treatment and control.
Proportion of subjects who experience rebleeding following initial hemostasis that requires subsequent medical intervention to re-achieve hemostasis within 24, 48, and 72 hours after the start of treatment | 72 hours following start of treatment
  Summarized as the proportion of subjects that met criteria and compared between active treatment and control.
Number of rebleeding episodes following initial hemostasis that require subsequent medical intervention to re-achieve hemostasis within 24, 48, and 72 hours after the start of treatment | 72 hours following start of treatment
  Summarized as the number of episodes per subject compared between active treatment and control.
Time to achieve hemostasis (in minutes) following the start of treatment in subjects with a bleed time of at least 10 minutes in either treatment period | 72 hours following start of treatment
  Time (in minutes) to achieve hemostasis will be compared between active treatment and control.
Proportion of subjects who experience adverse events including adverse skin reactions and other clinically significant findings on physical exam; clinically significant lab values; and clinically significant changes in vital signs. | 9 days
  Summarized as the proportion of subjects reporting adverse events compared between active treatment and control.
Systolic blood pressure | 7 days
  Summarized as observed values and change from baseline compared between active treatment and control.
Diastolic blood pressure | 7 days
  Summarized as observed values and change from baseline compared between active treatment and control.

CONTACTS AND LOCATIONS:
Locations (1):
- Accel Research Sites Network - DeLand, DeLand, Florida, United States

IPD SHARING:
Plan to Share IPD: No